CLINICAL TRIAL: NCT05189015
Title: Effect of Olmesartan or Amlodipine on Serum Angiotensin(1-7) Levels and Vascular Functions in Patients With Type 2 Diabetes and Hypertension
Brief Title: Effect of Olmesartan on Angiotensin(1-7) Levels and Vascular Functions in Diabetes and Hypertension
Acronym: Ang(1-7)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-1608-359-005
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Angiotensin/Renin/Aldosterone Hypertension; Hypertension; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2 | interventions — olmesartan; Olmesartan Medoxomil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olmesartan (Experimental): - Olmesartan group: Olmesartan, 20 (40) mg once a day, oral administration
  Interventions: Drug: Olmesartan
- Amlodipine (Active Comparator): - Comparator group: Amlodipine, 5 (10) mg once a day, oral administration
  Interventions: Drug: Olmesartan

INTERVENTIONS:
Drug: Olmesartan — - Olmesartan group: Olmesartan, 20 (40) mg once a day, oral administration
  Other Names: Olmesartan medoxomil

SUMMARY:
In this study, we will assess the change of serum ACE-2, angiotensin(1-7), and vascular function after using olmesartan (an ARB), compared to conventional anti-hypertensive drug, amlodipine in hypertensive patients with T2DM.

DETAILED DESCRIPTION:
Both ACE inhibitor and ARB produce inhibition of the renin-angiotensin system, so clinicians have regarded ACE inhibitor and ARB as effectively equivalent, including blood pressure lowering, improvement of congestive heart failure symptoms, inhibition of diabetic renal disease, reduction in stroke rates, and likely the prevention of new onset of diabetes mellitus. For an example, Ongoing Telmisartan Alone and in combination with Ramipril Global Endpoint Trial (ONTARGET) trial suggested that treatment with telmisartan or Ramipril reduces the cardiovascular outcomes to similar extent in patients with vascular disease or high-risk diabetes [2]. However, despite the similarities in mechanisms of two drugs, several recent meta-analysis showed the difference in treatment effect between ACE inhibitors and ARBs in patients with high risk of cardiovascular events, and it has become clear that these two classes of medication have significant differences with regard to their pharmacological properties and their molecular/cellular profiles [3, 4].

ACE inhibitors block angiotensin II synthesis form its precursor angiotensin I. However, ARBs block AT1 receptor, and hence ultimately angiotensin II is increased by a feedback mechanism. Although the cumulative effects of angiotensin II is not clearly elucidated yet, recent studies have established a new regulatory axis in the renin-angiotensin system (RAS). In this axis, angiotensin(1-7) is finally produced from Angiotensin I or Angiotensin II by the catalytic activity of angiotensin-converting enzyme 2 (ACE-2).

Diabetes mellitus is one of the leading risk factors for atherosclerosis and its complications including heart attacks and strokes. In addition, mortality rates are higher in diabetic than in non-diabetic patients [7]. The reason of cardiovascular risk in diabetes is not only related to hyperglycemia, but also commonly shares the risk factors such as hypertension, dyslipidemia, obesity, which are the characteristics of metabolic syndrome including insulin resistance and atherosclerosis. Atherosclerosis is an inflammatory disease that is related to low density lipoprotein, hypertension, diabetes, vascular inflammation, reactive oxygen species (ROS), and endothelial dysfunction. Angiotensin II makes an important role in this process and inflammatory cytokines such as IL-1, IL-6, TNF-α contribute as mediators.

Several clinical trials aimed at studying the benefits of RAS blockade in the diabetic complications. HOPE, RENAAL, IRMA2, IDNT, ONTARGET studies proved that ACE inhibitors or ARBs reduced the risk of diabetic complications [2, 8-11].

Recent studies proved that olmesartan, one of the ARBs, increases the activity of ACE-2 and angiotensin(1-7) level [12, 13]. 101 control subjects on no medication and 100 hypertensive patients treated with antihypertensive agents, including the calcium channel blockers, ACE inhibitor enalapril, and the angiotensin II receptor blockers losartan, candesartan, valsartan, telmisartan, and olmesartan, for more than 1 year were enrolled, and urinary ACE-2 level was measured. The result showed that urinary ACE-2 level was higher in the olmesartan-treated group, but not the other treatment groups, than in the control group. In addition, by multivariable regression analysis after adjustment of age, sex, and the correlated indices showed that the olmesartan was an independent predictor of urinary ACE-2 level [12]. The other study with 3 month old mice given olmesartan or hydralazine for 2 months revealed that olmesartan treatment inhibits cardiac hypertrophy independently of blood pressure not only through its AT1R blockade but partly through enhancement of ACE-2/angiotensin(1-7) [13]. However, there are some limitations. The former one was animal experiment, However, since they used many different drugs, the actual number of participants was quite small.

Therefore, understanding the change in concentration of serum ACE, ACE-2, angiotensin(1-7), and angiotensin-II should help clinicians select more appropriate drug between ACE inhibitors and ARBs with clear evidence. Moreover, since RAS antagonists are the first-line drugs for antihypertensive therapy in patients with T2DM, it is meaningful to understand the change of RAS-related factors in serum after using the drugs.

In this study, we will assess the change of serum ACE-2, angiotensin(1-7), and vascular function after using olmesartan (an ARB), compared to conventional anti-hypertensive drug, amlodipine in hypertensive patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 30 years old
* Type 2 diabetes by American Diabetes Association criteria
* HbA1c: 6.5% ≤ - < 10.0%
* Systolic blood pressure: 140 ≤ - < 180 mmHg or Diastolic blood pressure: 85 ≤ - < 110 mmHg
* Statin (-) or no change in low to moderate intensity statin [14] dose in recent 3 months

Exclusion Criteria:

* Contraindication of olmesartan or amlodipine
* History of RAS inhibitors (ACE inhibitors or ARBs) or calcium channel blockers in the previous 3 months
* Pregnant women, women with potential of pregnancy not using adequate contraception method as evaluated by the investigator, lactating women
* Type 1 diabetes or diabetes secondary to chronic pancreatitis or to pancreatectomy
* Confirmed cardiovascular disease (acute coronary syndrome, stroke, or transient ischemic attack) within 3 months of screening
* Chronic hepatitis B or C (except healthy carrier of HBV), liver disease (AST/ALT > 3-fold the upper limit of normal)
* Chronic kidney disease (serum creatinine > 2.0 mg/dL)
* Hyperkalemia serum potassium >5.0 mEq/L
* Any previous cancer within 5 years (except squamous cell cancer, cervical cancer, thyroid cancer with appropriate treatment) except thyroid cancer or carcinoma in situ

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
angiotensin(1-7) | 24 weeks
  Changes of serum angiotensin(1-7) at week 24 from baseline

SECONDARY OUTCOMES:
Blood pressure | 24 weeks
  Change in blood pressure from baseline to week 24
ACE-2 | 24 weeks
  Changes of serum ACE-2 at week 24 from baseline
Renin | 24 weeks
  Changes of serum renin at week 24 from baseline
Aldosterone | 24 weeks
  Changes of serum aldosterone at week 24 from baseline
hsCRP | 24 weeks
  Changes of serum hsCRP at week 24 from baseline
HbA1c | 24 weeks
  Change in HbA1c from baseline to week 24
glucose | 24 weeks
  Change in fasting glucose from baseline to week 24
Insulin | 24 weeks
  Change in fasting insulin from baseline to week 24
FMD | 24 weeks
  Change in flow mediated vasodilatation (FMD) from baseline to week 24
Microcirculation | 24 weeks
  Change in microcirculation from baseline to week 24
TG | 24 weeks
  Change in triglycerides from baseline to week 24
HDL | 24 weeks
  Change in HDL cholesterol from baseline to week 24
LDL | 24 weeks
  Change in LDL cholesterol from baseline to week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786
- [Derived] Kim K, Moon JH, Ahn CH, Lim S. Effect of olmesartan and amlodipine on serum angiotensin-(1-7) levels and kidney and vascular function in patients with type 2 diabetes and hypertension. Diabetol Metab Syndr. 2023 Mar 11;15(1):43. doi: 10.1186/s13098-023-00987-1. PMID 36899369